CLINICAL TRIAL: NCT03335033
Title: New Technologies to Determine Carotid Plaque Vulnerability: A Pilot Study to Assess Contrast-Enhanced Ultrasound (CEUS) and Shear Wave Elastography (SWE) in Patients With Significant Carotid Plaques
Brief Title: New Technologies to Determine Carotid Plaque Vulnerability in Patients With Significant Carotid Plaques
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew W. Urban, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17-001863
Record Dates: First submitted 2017-10-04; First posted 2017-11-07 (Actual); Results first posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Carotid Artery Plaque
Keywords: Carotid Plaque; Contrast Enhanced Ultrasound; Shear Wave Elastography; Endarterectomy; Stenosis
MeSH Terms: conditions — Carotid Stenosis; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Carotid Plaques with >70% Stenosis (Active Comparator): Subjects being seen in the Mayo Clinic Gonda Vascular Center who have a plaque causing a > 70% stenosis will be approached for recruitment to receive an ultrasound examination including duplex imaging, shear wave elastography and contrast-enhanced ultrasound.
  Interventions: Combination Product: Contrast-enhanced ultrasound; Device: Shear Wave Elastography; Device: Ultrasound Examination
- Carotid Plaques with 50-69% Stenosis (Active Comparator): Cardiovascular high-risk patients with moderate (50-69% diameter) stenosis carotid plaques from the Mayo Clinic Gonda Vascular Center will be approached for recruitment to receive an ultrasound examination including duplex imaging, shear wave elastography and contrast-enhanced ultrasound.
  Interventions: Combination Product: Contrast-enhanced ultrasound; Device: Shear Wave Elastography; Device: Ultrasound Examination

INTERVENTIONS:
Combination Product: Contrast-enhanced ultrasound — Subjects will receive a low mechanical index (0.17-0.20) imaging during ultrasound contrast agent intravenous infusion. Real-time cine-loop including longitudinal and transverse images obtained at least 3 seconds before and 5 minutes after the appearance of the contrast effect in the lumen of the carotid artery will be acquired and digitally stored for offline analysis. Also use of a 3D ultrasound transducer to evaluate the feasibility of using US images with contrast to assess the residual diameter of the diseased vessel. Specifically, two 3D acquisitions of each lesion would be obtained after contrast has been injected.
  Other Names: Lumason
Device: Shear Wave Elastography — Shear wave elastography will be performed with the General Electric Logiq E9 scanner acquiring images of each plaque in the longitudinal and transverse imaging planes. In each plane 10 measurements will be made and the in-phase/quadrature (IQ) data will be saved for further analysis. The plaque area in the imaging plane will be user-defined to extract the wave velocity values for a ROI analysis.
Device: Ultrasound Examination — A standard carotid US examination using Duplex imaging will performed using a linear array transducer to obtain longitudinal and transverse images. All ultrasound measurements will be made by a trained registered vascular technologist. Severity of stenosis of the plaque will be measured based on established protocol and guidelines.

SUMMARY:
The researchers are trying to determine if the characterization of "vulnerable" carotid artery plaques can be accomplished with ultrasound-based methods that look for vessels in the plaque and measure the plaque stiffness.

DETAILED DESCRIPTION:
All participants will receive a one time Carotid contrast-enhanced Ultrasound (CEUS) examination that may take 30-60 minutes. Follow up calls will be made to the Participants at 6, 12 ,24 and 36 months to ask about occurrence of major adverse cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Subject has carotid plaque with > 50% stenosis
* Subject is able to understand the study procedure and provide informed consent

Exclusion Criteria:

* Subject is pregnant or breast feeding
* Subject is unable to provide informed consent
* Subject has contraindication to the use of the Lumason contrast agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Urban, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Carotid Plaques With >70% Stenosis: Subjects who had a plaque causing a > 70% stenosis were approached for recruitment to receive an ultrasound examination including duplex imaging, shear wave elastography and contrast-enhanced ultrasound.
  Contrast-enhanced ultrasound: Subjects received a low mechanical index (0.17-0.20) imaging during ultrasound contrast agent intravenous infusion. Real-time cine-loop including longitudinal and transverse images obtained at least 3 seconds before and 5 minutes after the appearance of the contrast effect in the lumen of the carotid artery will be acquired and digitally stored for offline analysis. Also, use of a 3D ultrasound transducer to evaluate the feasibility of using US images with contrast to assess the residual diameter of the diseased vessel. Specifically, two 3D acquisitions of each lesion would be obtained after contrast has been injected.
  Shear Wave Elastography: Shear wave elastography as performed with the General Electric Logiq E9 scanner acquiring images of each plaque in the longitudinal and transverse imaging planes.
  Ultrasound Examination: A standard carotid US examination using Duplex imaging was performed using a linear array transducer to obtain longitudinal and transverse images. Severity of stenosis of the plaque will be measured based on established protocol and guidelines.
- Carotid Plaques With 50-69% Stenosis: Subjects with moderate (50-69% diameter) stenosis carotid plaques were approached for recruitment to receive an ultrasound examination including duplex imaging, shear wave elastography and contrast-enhanced ultrasound.
  Contrast-enhanced ultrasound: Subjects received a low mechanical index (0.17-0.20) imaging during ultrasound contrast agent intravenous infusion. Real-time cine-loop including longitudinal and transverse images obtained at least 3 seconds before and 5 minutes after the appearance of the contrast effect in the lumen of the carotid artery will be acquired and digitally stored for offline analysis. Also, use of a 3D ultrasound transducer to evaluate the feasibility of using US images with contrast to assess the residual diameter of the diseased vessel. Specifically, two 3D acquisitions of each lesion would be obtained after contrast has been injected.
  Shear Wave Elastography: Shear wave elastography as performed with the General Electric Logiq E9 scanner acquiring images of each plaque in the longitudinal and transverse imaging planes.
  Ultrasound Examination: A standard carotid US examination using Duplex imaging was performed using a linear array transducer to obtain longitudinal and transverse images. Severity of stenosis of the plaque will be measured based on established protocol and guidelines.
Period: Overall Study
Arm/Group | Carotid Plaques With >70% Stenosis | Carotid Plaques With 50-69% Stenosis
Started | 17 | 37
Completed | 17 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carotid Plaques With >70% Stenosis | Carotid Plaques With 50-69% Stenosis | Total
Number analyzed (Participants) | 17 | 37 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.4 (8.2) | 76.5 (7.6) | 76.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 14 | 21
  Male | 10 | 23 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 36 | 53
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 37 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 37 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Completed All of the Ultrasound Examinations
Description: Total number of subjects who completed all of the ultrasound examinations to determine visualization of arterial wall (contrast-enhanced ultrasound, 3-D volume ultrasound) and its mechanical properties (shear wave elastography).
Time Frame: 1 year after recruitment
Measure: Count of Participants; unit: Participants
Arm/Group | Carotid Plaques With >70% Stenosis | Carotid Plaques With 50-69% Stenosis
Number analyzed (Participants) | 17 | 37
Participants | 17 | 37

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 36 months
Arm/Group | Carotid Plaques With >70% Stenosis | Carotid Plaques With 50-69% Stenosis
All-Cause Mortality (participants affected / at risk) | 2/17 | 6/37
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/37
Other Adverse Events (participants affected / at risk) | 0/17 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT03335033/Prot_SAP_000.pdf